CLINICAL TRIAL: NCT06109805
Title: Identification and Multicentral Clinical Validation of Plasma Diagnostic Biomarkers for Gastric Cancer Based on Wide-targeted and Targeted Metabolomics
Brief Title: Plasma Metabolic Biomarkers for Gastric Cancer Diagnosis
Status: Completed | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Min Li, Deputy Director of Science and Technology Department, Beijing Friendship Hospital
Other Study IDs: BFHHZML20230010
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Only metabolites will be detected and analyzed in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Gastric cancer group: Patients diagnosed with gastric cancer, including early gastric cancer and advanced gastric cancer
  Interventions: Other: Gastric cancer
- Non-gastric cancer group: Patients diagnosed with benign gastric diseases or healthy controls

INTERVENTIONS:
Other: Gastric cancer — Patients diagnosed with gastric cancer, including early gastric cancer and advanced gastric cancer
  Groups: Gastric cancer group

SUMMARY:
The aim of this observational study is to comprehensively analyze the metabolites in plasma samples from gastric cancer patients using advanced mass spectrometry detection technology, in conjunction with both broad-spectrum and targeted metabolomics approaches. The goal is to construct a dedicated plasma metabolite database for gastric cancer patients. Simultaneously, we will delve into the exploration and validation of a series of metabolic biomarkers for early gastric cancer diagnosis. The objective is to establish a safer, more convenient, and more sensitive early screening method, thereby providing a reliable scientific foundation and critical evidence for improving the early diagnostic process for individuals at high risk of gastric cancer.

DETAILED DESCRIPTION:
Firstly, a wide-targeted metabolomic measurement will be conducted on plasma samples from the discovery cohort to identify potential metabolite candidate markers and construct a gastric cancer patient-specific metabolite database with extensive metabolite information.

Secondly, a more precise targeted metabolomic measurement will be conducted in the modeling cohort. Bioinformatics methods will be used to conduct an in-depth analysis of a wide range of metabolite information to screen out metabolic marker combinations with high gastric cancer-specific diagnostic efficacy.

Ultimately, an external validation cohort will be introduced to validate these metabolic biomarkers, aiming to ensure reliability and stability across different patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of gastric cancer or benign gastric diseases through gastroscopy and pathological examination.
* Collection of plasma samples prior to surgical treatment.
* Availability of complete clinical data.

Exclusion Criteria:

* Previous reception of anti-tumor treatments (including radiotherapy, chemotherapy, etc.) before blood collection.
* Coexistence of other systemic tumors.
* Absence of plasma sample collection before surgical treatment.
* Incomplete clinical data.
* Pregnancy status.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population included a range of subjects with gastric and non-gastric cancer, including patients with benign gastric disease and healthy controls, who were admitted to the main study center and other collaborating sub-center hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 1706 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Plasma metabolite content | Before receiving treatment for gastric cancer
  The outcome will be tested by metabolomics detection technology based on mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Li Min, Ph.D., Principal Investigator — Beijing Friendship Hospital
Locations (4):
- China (4):
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Renmin Hospital of Wuhan University, Wuhan
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan

IPD SHARING:
Plan to Share IPD: No